CLINICAL TRIAL: NCT02758015
Title: Countering the Gastric ph Effect of a Standardized Meal in Healthy Volunteers Using Clinical Doses of Betaine Hydrochloride
Brief Title: Effect of Betaine and Food on Gastric pH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16-18635
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Healthy
Keywords: betaine; betaine hydrochloride; healthy volunteer; gastric pH
MeSH Terms: interventions — Betaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standardized Meal (Active Comparator): Standardized meal given to patients.
  Interventions: Other: Standardized Meal
- Beatine PO (by mouth) 1500mg (Experimental): Betaine (natural supplement)
  Interventions: Other: Standardized Meal; Dietary Supplement: Betaine Hydrochloride 1500mg
- Betaine PO (by mouth) 3000mg (Experimental): Betaine (natural supplement)
  Interventions: Other: Standardized Meal; Dietary Supplement: Betaine Hydrochloride 3000mg
- Betaine PO (by mouth) 4500mg (Experimental): Betaine (natural supplement)
  Interventions: Other: Standardized Meal; Dietary Supplement: Betaine Hydrochloride 4500mg

INTERVENTIONS:
Other: Standardized Meal
Dietary Supplement: Betaine Hydrochloride 1500mg — Betaine hydrochloride (natural supplement) administered after standardized meal.
  Arms: Beatine PO (by mouth) 1500mg
Dietary Supplement: Betaine Hydrochloride 3000mg — Betaine hydrochloride (natural supplement) administered after standardized meal.
  Arms: Betaine PO (by mouth) 3000mg
Dietary Supplement: Betaine Hydrochloride 4500mg — Betaine hydrochloride (natural supplement) administered after standardized meal.
  Arms: Betaine PO (by mouth) 4500mg

SUMMARY:
Food will decrease stomach acidity due to its buffering effect.This has implications when providing drugs that are dosed with food but require higher levels of stomach acid, such as some medications commonly used for HIV patients. This study will attempt to determine the dose of betaine hydrochloride (over the counter acid supplement) at which the effect of food on stomach acid could be countered. Additionally, this study will evaluate the ability of a natural supplement (betaine hydrochloride) to affect the gastric pH following a standardized meal in healthy volunteers. The investigators predict that 4500mg of betaine hydrochloride will have the greatest effect on gastric pH.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-64 years of age;
* Healthy adult with no active medical problems or significant chronic diseases as determined by the study doctor based on history, physical exam;
* BMI between 18.5 - 32 kg/m2;
* Taking no medications 2 weeks before and during the study enrollment, including drugs of abuse, prescription or OTC medications (except acetaminophen);
* Be able to provide written informed consent and comply with requirements of the study;
* Avoid eating grapefruit and drinking grapefruit juice from 7 days before the first study day until completion of the entire study;
* Abstinence from alcoholic beverages, caffeinated beverages and orange juice from 3pm the night before a study day until completion of that study day;
* Fast from food and beverages at least 8 hours prior to the study day;
* Be able to read, speak and understand English

Exclusion Criteria:

* Subjects with a history of gastrointestinal disease including gastroesophageal reflux disease, gastritis, peptic ulcer disease or dyspepsia.
* Subjects with a fasting gastric pH of > 4 (i.e. hypochlorhydria)
* Subjects with history of dysphagia, achalasia, or difficulty swallowing capsules, tablets or pills.
* Subjects on prescription or chronic over-the counter medications (including hormonal contraceptives);
* Subjects with liver failure or LFTs >2x upper limit of normal;
* Subjects with clinically significant elevations in SCr, BUN or other screening laboratory tests as determined by study physician;
* Subjects with Hct < 30 mg/dL, WBC < 2000/μL, ANC < 1000/μL, or platelet count < 150,000/μL;
* Subjects with a history or presence of an abnormal ECG, including demonstration of a baseline corrected Fridericia's QT interval (QTcF) >450ms, which in the opinion of the study physician, is clinically significant;
* Subjects who smoke tobacco;
* Subjects with ongoing alcohol or illegal drug use;
* Subjects who are pregnant, lactating or attempting to conceive;
* Subjects unable to follow protocol instructions or protocol criteria.
* Anyone who in the opinion of the study investigators is unable to participate in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2016-06; Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Change in Gastric pH After Administration of Standardized Meal | 15 minutes
  After Heidelberg capsule is placed and baseline gastric levels have been recorded using the Heidelberg Capsule (HC), which sends real-time signals to a computer system that visually plots intestinal pH on a minute-by-minute basis, a standardized meal is given. Gastric pH is measured for 15 minutes after the administration of the meal.
Change in Gastric pH After Administration of Standardized Meal and Betaine hydrochloride | 3 hours
  After 15 minutes of gastric pH monitoring following the standardized meal, betaine hydrochloride will be administered and its effect on the ability to mitigate that rise in gastric pH will be determined using the Heidelberg capsule over the span of approximately 3 hours. This will be done three separate times with 3 doses (1500mg, 3000mg, and 4500mg) dosed orally with 90ml of water.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Z Benet, PhD, Principal Investigator — University of California, San Francisco; Lynda A Frassetto, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Clinical Research Center, UCSF, San Francisco, California, United States

REFERENCES:
- [Derived] Surofchy DD, Frassetto LA, Benet LZ. Food, Acid Supplementation and Drug Absorption - a Complicated Gastric Mix: a Randomized Control Trial. Pharm Res. 2019 Sep 4;36(11):155. doi: 10.1007/s11095-019-2693-5. PMID 31485804